CLINICAL TRIAL: NCT01277367
Title: A Prospective, Randomized Clinical Trial Comparing the Effectiveness of Different Types of Incentives in Increasing Physical Activity Behavior on the Vitality Health Promotion Programme
Brief Title: Vitality Health Incentives for Physical Activity
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 811570
Record Dates: First submitted 2011-01-12; First posted 2011-01-14 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Obesity
Keywords: Obesity; Sedentary; Physical activity; exercise; incentives
MeSH Terms: conditions — Obesity; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- A (Active Comparator): These members will be offered no additional incentives
  Interventions: Behavioral: Discovery Vitality base program
- B (Experimental): These members will receive regular communications by Discovery Vitality.
  Interventions: Behavioral: Discovery Vitality base program; Behavioral: Communication
- C (Experimental): These members will nominate a charity which will benefit financially based on participants' level of physical activity.
  Interventions: Behavioral: Discovery Vitality base program; Behavioral: Charitable Incentive
- D (Experimental): These members are entered into a prize draw for a monthly cash prize if they achieve physical activity targets.
  Interventions: Behavioral: Discovery Vitality base program; Behavioral: Prize Draw Incentive
- E (Experimental): These members will receive a direct payment.
  Interventions: Behavioral: Discovery Vitality base program; Behavioral: Direct Payment
- F (Experimental): These members will be offered the opportunity to choose one of three incentive options at the time of enrollment in the study.
  Interventions: Behavioral: Discovery Vitality base program; Behavioral: Free Choice

INTERVENTIONS:
Behavioral: Discovery Vitality base program — The existing Discovery Vitality health promotion base program, which offers points for various levels of physical activity.
Behavioral: Communication — Participants will be sent regular communications by Discovery Vitality -equivalent to the level of communications in the other incentive groups - which will provide information and tips about ways of accumulating Vitality points on the existing programme (concerning fitness-related activities, in particular).
  Arms: B
Behavioral: Charitable Incentive — Members will be asked to nominate a charity, from a selection of charities, which will benefit financially (Discovery Vitality will make a direct payment to a nominated charity) based on their (member's) level of participation in points-earning physical activity. Individuals will receive one of four possible payouts, corresponding to their level of engagement, for their selected charity (amounts given below). In addition, members will be sent regular updates of activities by their nominated charities (This will be operationalised and facilitated by Vitality- and as such, no direct mailing from nominated charity will take place, to maintain confidentiality.)
  Arms: C
Behavioral: Prize Draw Incentive — Members will be entered into a prize draw for a monthly cash-prize if they achieve physical activity targets. Four lottery payouts, corresponding to their levels of engagement, will be made on a monthly basis. All members will be sent information regarding the winnings of those that are drawn (unlinked to personal identifiers, but to motivate).
  Arms: D
Behavioral: Direct Payment — Members will receive a direct payment (in the form of gift voucher) of one of four possible amounts depending on the level of participation in fitness-related activities equivalent in expected value to the payouts in arms 3 and 4.
  Arms: E
Behavioral: Free Choice — Members will be asked to choose one of the three aforementioned incentive options on enrollment to the study.
  Arms: F

SUMMARY:
The aim of the study is to prospectively compare the effectiveness of diverse incentives on physical activity behaviour, in a cohort of newly-enrolled, adult members of the Vitality health promotion programme based in South Africa.

DETAILED DESCRIPTION:
Newly enrolled adult members of the Discovery Health medical plan who have, themselves, prospectively registered for the Vitality health promotion programme will be eligible for the study, and will be invited to participate by Discovery Vitality. A final sample of 9000 adult members, who are recruited and have agreed to participate, will be randomly allocated by Discovery Vitality (with replacement) to one of six study (incentive) groups (n=1500 per group) and followed for six months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* enrolled in Vitality

Exclusion Criteria:

* under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Engagement in physical activity | 6 months
  Levels of engagement in fitness related activities as measured by 1) continuous measure of Vitality fitness program points accrued, and 2) frequency count or proportion of members by fitness level groups

SECONDARY OUTCOMES:
Fitness points earned | 6 months
  The standard Vitality program offers members the ability to accumulate points for physical activity behavior through various means.
Gym visits | 6 months
  Average number of gym visits over the six month period will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Patel, MD, Study Chair — Discovery Holdings, LTD
Locations (4):
- United States (2):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Carnegie Mellon University, Pittsburgh, Pennsylvania
- South Africa (2):
  - University of Cape Town, Cape Town
  - Discovery Vitality, Johannesburg